CLINICAL TRIAL: NCT01326702
Title: A Phase 1b/2a Study of ABT-888 in Combination With Bendamustine +/- Rituximab in Lymphoma, Multiple Myeloma and Solid Tumors
Brief Title: Veliparib, Bendamustine Hydrochloride, and Rituximab in Treating Patients With Relapsed or Refractory Lymphoma, Multiple Myeloma, or Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02583; NCI-2011-02583 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000697580; 10-174 (Other: Memorial Sloan-Kettering Cancer Center); 8818 (Other: CTEP); P30CA008748 (NIH); U01CA069856 (NIH)
Record Dates: First submitted 2011-03-30; First posted 2011-03-31 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-11

CONDITIONS: Adult B Acute Lymphoblastic Leukemia; Adult Nasal Type Extranodal NK/T-Cell Lymphoma; Adult Solid Neoplasm; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-Cell Lymphoma; Chronic Lymphocytic Leukemia; Cutaneous B-Cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Hepatosplenic T-Cell Lymphoma; Intraocular Lymphoma; Lymphomatous Involvement of Non-Cutaneous Extranodal Site; Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Nodal Marginal Zone Lymphoma; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-Cell Leukemia/Lymphoma; Recurrent Cutaneous T-Cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides and Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Plasma Cell Myeloma; Small Intestinal Lymphoma; Splenic Marginal Zone Lymphoma; Testicular Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Intraocular Lymphoma; Lymphoma, T-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Hairy Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Bendamustine Hydrochloride; Rituximab; veliparib

ARMS (1):
- Treatment (veliparib, bendamustine hydrochloride, rituximab) (Experimental): Patients receive veliparib PO BID on days 1-7 and bendamustine hydrochloride IV over 30-60 minutes on days 1-2. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Once the maximum-tolerated dose is determined, a cohort of patients receives veliparib and bendamustine hydrochloride as above and rituximab IV on day 1. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bendamustine Hydrochloride; Other: Pharmacological Study; Biological: Rituximab; Drug: Veliparib

INTERVENTIONS:
Drug: Bendamustine Hydrochloride — Given IV
  Other Names: Bendamustin Hydrochloride; Cytostasan Hydrochloride; Levact; Ribomustin; SyB L-0501; Treanda
Other: Pharmacological Study — Correlative studies
Biological: Rituximab — Given IV
  Other Names: BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar BI 695500; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; RTXM83
Drug: Veliparib — Given PO
  Other Names: ABT-888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase I/II trial studies the side effects and the best dose of veliparib when given together with bendamustine hydrochloride and rituximab and to see how well they work in treating patients with lymphoma, multiple myeloma, or solid tumors that have come back or have not responded to treatment. Veliparib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as bendamustine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some find cancer cells and help kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. Giving veliparib together with bendamustine hydrochloride and rituximab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum-tolerated dose (MTD) of ABT-888 (veliparib) in combination with bendamustine (bendamustine hydrochloride) in patients with solid tumors, lymphoma, or multiple myeloma. (Phase Ib) II. To establish the safety of ABT-888 in combination with bendamustine and rituximab in an expansion cohort of patients with non-Hodgkin lymphoma (NHL). (Phase Ib) III. To assess the toxicity profile of this regimen in the above patients. (Phase Ib) IV. To determine the complete response (CR) rate in patients with indolent NHL or mantle cell lymphoma (MCL) treated with ABT-888 + bendamustine + rituximab. (Phase IIa)

SECONDARY OBJECTIVES:

I. To assess response rates and survival parameters of patients treated with ABT-888 + bendamustine +/- rituximab. (Phase Ib) II. To assess pharmacokinetic parameters of ABT-888 in this regimen. (Phase Ib) III. To assess progression-free survival, overall survival, and duration of remission of patients with indolent NHL and MCL treated with ABT-888 + bendamustine + rituximab. (Phase IIa)

OUTLINE: This is a phase I, dose-escalation study of veliparib followed by a phase II study.

Patients receive veliparib orally (PO) twice daily (BID) on days 1-7 and bendamustine hydrochloride intravenously (IV) over 30-60 minutes on days 1-2. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Once the maximum-tolerated dose is determined, a cohort of patients receives veliparib and bendamustine hydrochloride as above and rituximab IV on day 1. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1b: Patients must have a histologically confirmed solid malignancy, lymphoma or multiple myeloma for which standard curative or palliative measures do not exist, are no longer effective, or for which the patient is not eligible or refuses; phase 1b cohort expansion: patients must have a histologically confirmed cluster of differentiation (CD)-20 positive B-cell non-Hodgkin lymphoma for which standard curative or palliative measures do not exist, are no longer effective, or for which the patient is not eligible or refuses; phase 2a: patients must have histologically or cytologically confirmed marginal zone B-cell lymphoma, small lymphocytic lymphoma, lymphoplasmacytic lymphoma or mantle cell lymphoma, and must have at least one measureable site of disease
* For lymphoma and multiple myeloma patients: patients who have relapsed or are refractory to at least one prior chemotherapeutic regimen or biologic agent; patients must either be ineligible for or have refused curative options for treatment, including stem cell transplant, if applicable
* For solid tumor patients: relapsed or refractory to at least one prior chemotherapeutic regimen or biologic agent; patients must either be ineligible for or have refused curative options for treatment
* Patients must have had a rest period of at least 3 weeks since prior chemotherapy or radiation therapy, 6 weeks if the last regimen included carmustine (BCNU) or mitomycin C; there must be a rest period of at least 3 months if the last therapy was immunotherapy or radioimmunotherapy (unless the disease has progressed since treatment)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Absolute neutrophil count (ANC) >= 1,000/mcL
* Platelets >= 100,000/mcL unsupported by transfusion within the prior 2 weeks
* Hemoglobin >= 8.0 g/dL unsupported by transfusion within the prior 2 weeks
* Total bilirubin =< 2 x upper normal institutional limits; in patients with Gilbert's disease or documented liver metastases, total bilirubin up to 3 x upper limits of normal (ULN) will be allowed
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min for patients with creatinine levels above institutional normal
* Patients with prior stem cell transplant will be eligible as long as they have not relapsed or progressed within 100 days post-transplant and they meet the above inclusion criteria
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal, barrier method of birth control, or abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Toxicities from prior therapies must have resolved to baseline, or be =< grade 2 and stable for at least one month
* Patient must be able to swallow pills
* Patients with central nervous system (CNS) metastases must be stable after therapy for > 3 months and off steroid treatment prior to study enrollment

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered to baseline (or are not at stable grade =< 2) from adverse events due to agents administered more than 3 weeks earlier; patients who have received immunotherapy or radioimmunotherapy within 3 months, unless disease has progressed since treatment; patients who have been administered ABT-888 as part of a single or limited dosing study, such as a phase 0 study, will not be excluded from participating in this study solely because of receiving prior ABT-888
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ABT-888, bendamustine or mannitol; patients enrolling in the cohort expansion or phase 2 portions of the study who have been intolerant of repeated doses of rituximab in the past will be excluded (patients who have had infusion reactions to their initial dose of rituximab will not be excluded)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with ABT-888
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are eligible if their HIV is under adequate control with an antiretroviral regimen that has been stable for >= 4 weeks, as long as the CD4 count is > 300; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated; patients on zidovudine or stavudine would not be eligible
* Patients with active seizure or a history of seizure are not eligible
* Patients with uncontrolled CNS metastasis are not eligible
* Patients with unrelated prior malignancies must have undergone potentially curative therapy for their prior malignancy, have no evidence of that disease for three years, or be deemed at low risk for recurrence of their prior malignancy by her/his treating physician; patients with dermal squamous cell carcinoma, basal cell carcinoma or melanoma in situ that has been completely excised will be eligible following excision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Gerecitano, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Soumerai JD, Zelenetz AD, Moskowitz CH, Palomba ML, Hamlin PA Jr, Noy A, Straus DJ, Moskowitz AJ, Younes A, Matasar MJ, Horwitz SM, Portlock CS, Konner JA, Gounder MM, Hyman DM, Voss MH, Fury MG, Gajria D, Carvajal RD, Ho AL, Beumer JH, Kiesel B, Zhang Z, Chen A, Little RF, Jarjies C, Dang TO, France F, Mishra N, Gerecitano JF. The PARP Inhibitor Veliparib Can Be Safely Added to Bendamustine and Rituximab and Has Preliminary Evidence of Activity in B-Cell Lymphoma. Clin Cancer Res. 2017 Aug 1;23(15):4119-4126. doi: 10.1158/1078-0432.CCR-16-3068. Epub 2017 Mar 17. PMID 28314788

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1-Bendamustine 70 mg/m2, ABT-888 50 mg: Bendamustine 70 mg/m2, ABT-888 50 mg
- Dose Level 2: Bendamustine 90 mg/m2, ABT-888 50 mg: Bendamustine 90 mg/m2, ABT-888 50 mg
- Dose Level 3: Bendamustine 90 mg/m2, ABT-888 100 mg BID: Bendamustine 90 mg/m2, ABT-888 100 mg BID
- Dose Level 4: Bendamustine 90 mg/m2, ABT-888 150 mg BID: Bendamustine 90 mg/m2, ABT-888 150 mg BID
- Dose Level 5: Bendamustine 90 mg/m2, ABT-888 200 mg BID: Bendamustine 90 mg/m2, ABT-888 200 mg BID
- Dose Level 6: Bendamustine 90 mg/m2, ABT-888 300 mg BID: Bendamustine 90 mg/m2, ABT-888 300 mg BID
- Dose Level 7: Bendamustine 90 mg/m2, ABT-888 400 mg BID: Bendamustine 90 mg/m2, ABT-888 400 mg BID
Period: Overall Study
Arm/Group | Dose Level 1-Bendamustine 70 mg/m2, ABT-888 50 mg | Dose Level 2: Bendamustine 90 mg/m2, ABT-888 50 mg | Dose Level 3: Bendamustine 90 mg/m2, ABT-888 100 mg BID | Dose Level 4: Bendamustine 90 mg/m2, ABT-888 150 mg BID | Dose Level 5: Bendamustine 90 mg/m2, ABT-888 200 mg BID | Dose Level 6: Bendamustine 90 mg/m2, ABT-888 300 mg BID | Dose Level 7: Bendamustine 90 mg/m2, ABT-888 400 mg BID
Started | 3 | 3 | 6 | 4 | 5 | 15 | 7
Completed | 1 | 1 | 1 | 1 | 1 | 7 | 0
Not Completed | 2 | 2 | 5 | 3 | 4 | 8 | 7
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — progressive disease | 1 | 1 | 3 | 1 | 3 | 2 | 3
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 1 | 3
Not completed — Not Treated | 0 | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1: Bendamustine 70 mg/m2, ABT-888 50 mg: Dose Level 1: Bendamustine 70 mg/m2, ABT-888 50 mg
- Dose Level 2: Bendamustine 90 mg/m2, ABT-888 50 mg: Dose Level 2: Bendamustine 90 mg/m2, ABT-888 50 mg
- Dose Level 3: Bendamustine 90 mg/m2, ABT-888 100 mg BID: Dose Level 3: Bendamustine 90 mg/m2, ABT-888 100 mg BID
- Dose Level 4: Bendamustine 90 mg/m2, ABT-888 150 mg BID: Dose Level 4: Bendamustine 90 mg/m2, ABT-888 150 mg BID
- Dose Level 5: Bendamustine 90 mg/m2, ABT-888 200 mg BID: Dose Level 5: Bendamustine 90 mg/m2, ABT-888 200 mg BID
- Dose Level 6: Bendamustine 90 mg/m2, ABT-888 300 mg BID: Dose Level 6: Bendamustine 90 mg/m2, ABT-888 300 mg BID
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: Bendamustine 70 mg/m2, ABT-888 50 mg | Dose Level 2: Bendamustine 90 mg/m2, ABT-888 50 mg | Dose Level 3: Bendamustine 90 mg/m2, ABT-888 100 mg BID | Dose Level 4: Bendamustine 90 mg/m2, ABT-888 150 mg BID | Dose Level 5: Bendamustine 90 mg/m2, ABT-888 200 mg BID | Dose Level 6: Bendamustine 90 mg/m2, ABT-888 300 mg BID | Dose Level 7: Bendamustine 90 mg/m2, ABT-888 400 mg BID | Total
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 5 | 15 | 7 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 4 | 4 | 1 | 8 | 3 | 22
  >=65 years | 2 | 2 | 2 | 0 | 4 | 7 | 4 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 5 | 2 | 2 | 8 | 6 | 26
  Male | 2 | 1 | 1 | 2 | 3 | 7 | 1 | 17
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 4 | 5 | 15 | 7 | 43

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Veliparib When Combined With Bendamustine Hydrochloride
Description: Maximum Tolerated Dose (MTD) reflects the highest dose of Veliparib when combined with Bendamustine Hydrochloride that did not cause a DLT. The maximum tolerated dose (MTD) was defined as the highest dose level at which 33% of patients experienced DLT.
Time Frame: 28 days
Population: The MTD was established at Dose Level 6 Veliparib 300mg PO BID plus Bendamustine 90 mg/m2
Measure: Number; unit: mg
Groups:
- All Study Participants: All Study Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 43
mg | 300

2. Primary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI and/or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progression of Disease (POD); POD, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Complete Response (CR), Disappearance of all target lesions.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1-Bendamustine 70 mg/m2, ABT-888 50 mg | Dose Level 2: Bendamustine 90 mg/m2, ABT-888 50 mg | Dose Level 3: Bendamustine 90 mg/m2, ABT-888 100 mg BID | Dose Level 4: Bendamustine 90 mg/m2, ABT-888 150 mg BID | Dose Level 5: Bendamustine 90 mg/m2, ABT-888 200 mg BID | Dose Level 6: Bendamustine 90 mg/m2, ABT-888 300 mg BID | Dose Level 7: Bendamustine 90 mg/m2, ABT-888 400 mg BID
Number analyzed (Participants) | 3 | 3 | 5 | 2 | 3 | 14 | 2
Participants
  Complete Response | 0 | 0 | 1 | 0 | 0 | 4 | 0
  Partial Response | 1 | 1 | 0 | 0 | 1 | 4 | 0
  Stable Disease | 1 | 2 | 2 | 2 | 0 | 5 | 0
  Progression of Disease | 1 | 0 | 2 | 0 | 2 | 1 | 2

3. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse events assessed by NCI CTCAE version 4.0 (Phase Ib) See adverse events section.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Dose Level 1-Bendamustine 70 mg/m2, ABT-888 50 mg | Dose Level 2: Bendamustine 90 mg/m2, ABT-888 50 mg | Dose Level 3: Bendamustine 90 mg/m2, ABT-888 100 mg BID | Dose Level 4: Bendamustine 90 mg/m2, ABT-888 150 mg BID | Dose Level 5: Bendamustine 90 mg/m2, ABT-888 200 mg BID | Dose Level 6: Bendamustine 90 mg/m2, ABT-888 300 mg BID | Dose Level 7: Bendamustine 90 mg/m2, ABT-888 400 mg BID
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 5 | 15 | 7
participants | 3 | 3 | 4 | 2 | 2 | 5 | 3

4. Secondary Outcome: Complete Response (CR) to Study Treatment (Phase IIa)
Description: Summary statistics will be used for CR. Responses will be evaluated by the International Uniform Response Criteria for Multiple Myeloma.
Time Frame: 2 years
Population: Dose Level 7; Bendamustine 90mg/m2, ABT-888 400mg BID Participants treated on Dose Level 7 make up the cohort expansion of VBR in participants with CD20+ B-cell lymphoma.
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Participants | 5

5. Secondary Outcome: Duration of Remission (Phase IIa)
Time Frame: From the first documented response to the first documented progression or death, assessed up to 30 days post-treatment
Population: Data were not collected
Groups:
- Dose Level 1: Bendamustine 70 mg/m2, ABT-888 50 mg: Bendamustine 70 mg/m2, ABT-888 50 mg
Arm/Group | Dose Level 1: Bendamustine 70 mg/m2, ABT-888 50 mg | Dose Level 2: Bendamustine 90 mg/m2, ABT-888 50 mg | Dose Level 3: Bendamustine 90 mg/m2, ABT-888 100 mg BID | Dose Level 4: Bendamustine 90 mg/m2, ABT-888 150 mg BID | Dose Level 5: Bendamustine 90 mg/m2, ABT-888 200 mg BID | Dose Level 6: Bendamustine 90 mg/m2, ABT-888 300 mg BID | Dose Level 7: Bendamustine 90 mg/m2, ABT-888 400 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Overall Survival (Phase IIa)
Description: Kaplan-Meier estimates will be calculated and log-rank tests will be employed when certain comparisons are needed.
Time Frame: Up to 30 days post-treatment
Population: Data were not collected
Arm/Group | Dose Level 1-Bendamustine 70 mg/m2, ABT-888 50 mg | Dose Level 2: Bendamustine 90 mg/m2, ABT-888 50 mg | Dose Level 3: Bendamustine 90 mg/m2, ABT-888 100 mg BID | Dose Level 4: Bendamustine 90 mg/m2, ABT-888 150 mg BID | Dose Level 5: Bendamustine 90 mg/m2, ABT-888 200 mg BID | Dose Level 6: Bendamustine 90 mg/m2, ABT-888 300 mg BID | Dose Level 7: Bendamustine 90 mg/m2, ABT-888 400 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Pharmacokinetic Parameters of Veliparib (Phase Ib)
Description: Area Under the Curve from time zero to 12 hours following Veliparib administration
Time Frame: From time zero to 12 hours on day 2 of course 1
Measure: Geometric Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | Dose Level 1-Bendamustine 70 mg/m2, ABT-888 50 mg | Dose Level 2: Bendamustine 90 mg/m2, ABT-888 50 mg | Dose Level 3: Bendamustine 90 mg/m2, ABT-888 100 mg BID | Dose Level 4: Bendamustine 90 mg/m2, ABT-888 150 mg BID | Dose Level 5: Bendamustine 90 mg/m2, ABT-888 200 mg BID | Dose Level 6: Bendamustine 90 mg/m2, ABT-888 300 mg BID | Dose Level 7: Bendamustine 90 mg/m2, ABT-888 400 mg BID
Number analyzed (Participants) | 3 | 2 | 6 | 3 | 5 | 6 | 7
μg*h/mL | 1.79 (0.41) | 3.58 (0.93) | 7.93 (1.90) | 12.6 (3.8) | 16.9 (11.1) | 19.0 (10.5) | 25.0 (14.6)

8. Secondary Outcome: Progression-free Survival Using RECIST Version 1.1 (Phase IIa)
Description: Kaplan-Meier estimates will be calculated and log-rank tests will be employed when certain comparisons are needed. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.
Time Frame: 2 years
Population: Participants treated on Dose Level 7 make up the cohort expansion of VBR in participants with CD20+ B-cell lymphoma.
Measure: Median (Full Range); unit: Months
Groups:
- All Study Participants: Dose Level 7; Bendamustine 90mg/m2, ABT-888 400mg BID
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Months | 14.2 [2 to 20.1]

9. Secondary Outcome: Participants With Dose Limiting Toxicities
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | Dose Level 1-Bendamustine 70 mg/m2, ABT-888 50 mg | Dose Level 2: Bendamustine 90 mg/m2, ABT-888 50 mg | Dose Level 3: Bendamustine 90 mg/m2, ABT-888 100 mg BID | Dose Level 4: Bendamustine 90 mg/m2, ABT-888 150 mg BID | Dose Level 5: Bendamustine 90 mg/m2, ABT-888 200 mg BID | Dose Level 6: Bendamustine 90 mg/m2, ABT-888 300 mg BID | Dose Level 7: Bendamustine 90 mg/m2, ABT-888 400 mg BID
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 5 | 15 | 7
participants | 0 | 0 | 1 | 0 | 0 | 1 | 2

ADVERSE EVENTS:
Arm/Group | Dose Level 1: Bendamustine 70 mg/m2, ABT-888 50 mg | Dose Level 2: Bendamustine 90 mg/m2, ABT-888 50 mg | Dose Level 3: Bendamustine 90 mg/m2, ABT-888 100 mg BID | Dose Level 4: Bendamustine 90 mg/m2, ABT-888 150 mg BID | Dose Level 5: Bendamustine 90 mg/m2, ABT-888 200 mg BID | Dose Level 6: Bendamustine 90 mg/m2, ABT-888 300 mg BID | Dose Level 7: Bendamustine 90 mg/m2, ABT-888 400 mg BID
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 0/6 | 0/4 | 0/5 | 0/15 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/3 | 3/6 | 2/4 | 2/5 | 5/15 | 3/7
Other Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 1/6 | 0/4 | 0/5 | 0/15 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: Bendamustine 70 mg/m2, ABT-888 50 mg (N=3) | Dose Level 2: Bendamustine 90 mg/m2, ABT-888 50 mg (N=3) | Dose Level 3: Bendamustine 90 mg/m2, ABT-888 100 mg BID (N=6) | Dose Level 4: Bendamustine 90 mg/m2, ABT-888 150 mg BID (N=4) | Dose Level 5: Bendamustine 90 mg/m2, ABT-888 200 mg BID (N=5) | Dose Level 6: Bendamustine 90 mg/m2, ABT-888 300 mg BID (N=15) | Dose Level 7: Bendamustine 90 mg/m2, ABT-888 400 mg BID (N=7)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasms ben/mal/unk (in cyst/polyp) Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemolysis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: Bendamustine 70 mg/m2, ABT-888 50 mg (N=3) | Dose Level 2: Bendamustine 90 mg/m2, ABT-888 50 mg (N=3) | Dose Level 3: Bendamustine 90 mg/m2, ABT-888 100 mg BID (N=6) | Dose Level 4: Bendamustine 90 mg/m2, ABT-888 150 mg BID (N=4) | Dose Level 5: Bendamustine 90 mg/m2, ABT-888 200 mg BID (N=5) | Dose Level 6: Bendamustine 90 mg/m2, ABT-888 300 mg BID (N=15) | Dose Level 7: Bendamustine 90 mg/m2, ABT-888 400 mg BID (N=7)
Anemia (Blood and lymphatic system disorders) | 1 (8) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (5) | 1 (4) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less